CLINICAL TRIAL: NCT01322451
Title: A Randomized, Open Label, 2-way Crossover Study to Compare the Oral Bioavailability of 2 Solid Dose Formulations of GLPG0259 After Single-dose Intake in Healthy Subjects
Brief Title: Oral Bioavailability of Two Solid Formulations of GLPG0259.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Senior Vice President Development, Galapagos NV
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GLPG0259-CL-104; 2010-022456-23 (EudraCT Number)
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single oral dose, single capsule (Experimental)
  Interventions: Drug: GLPG0259 free base
- Single oral dose, two capsules (Experimental)
  Interventions: Drug: GLPG0259 fumarate

INTERVENTIONS:
Drug: GLPG0259 fumarate — single oral dose, two capsules each containing 25 mg of GLPG0259 fumarate
  Arms: Single oral dose, two capsules
Drug: GLPG0259 free base — single oral dose, GLPG0259, 50 mg solid formulation
  Arms: Single oral dose, single capsule

SUMMARY:
The purpose of the study is to evaluate the relative bioavailability of two solid oral formulations of GLPG0259 administered after a meal.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m², inclusive.

Exclusion Criteria:

* significantly abnormal platelet function or coagulopathy
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Bioavailability of two solid dosage formulations of GLPG0259 | up to 96 hours postdose

SECONDARY OUTCOMES:
Safety and tolerability of GLPG0259 | up to 96 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Johan Beetens, PharmD, PhD, Study Director — Galapagos NV; Lien Gheyle, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium